CLINICAL TRIAL: NCT01292850
Title: Skin Sterility After Ethyl-Chloride Spray
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Robin Gehrmann, M.D. Assistant Professor Department of Orthopaedics, Chief of Sports Medicine, New Jersey Medical School, UMDNJ
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0120080090
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Skin Sterility After Use of Ethyl-chloride Spray.
Keywords: Topical; Skin; sterility; ethylchloride; ethyl; chloride; spray
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers: 15 healthy volunteers were recruited

SUMMARY:
The aim of this study is to investigate sterility of ethyl-chloride topical anesthetic spray when used prior to an injection. The hypothesis is that the spray does not change the sterility of the injection site after skin is prepped.

DETAILED DESCRIPTION:
This is an IRB-approved, prospective, blinded, controlled study. In the first set of experiments, skin sterility is assessed. Healthy adult subjects are prepared for mock injections of shoulders and knees. No injection is performed. Each site has a set of 3 skin cultures: 1) prior to the alcohol prep (pre-prep), 2) post-alcohol prep (pre-spray), and 3) after ethyl-chloride was sprayed on the site (post-spray). In the second set of experiments, sterility of ethyl chloride is tested directly by culturing the liquid from the spray bottles.

ELIGIBILITY:
Inclusion Criteria:

* age -- 18-85
* healthy skin at shoulder and knee area

Exclusion Criteria:

* allergy to ethyl-chloride
* skin lesions at shoulder or knee

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healty adult (18-85) volunteers
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
culture positivity | 5 days
  Cultures before and after Ethyl-Chloride spray are compared to see if there is any difference.

SECONDARY OUTCOMES:
Native skin flora | 5days
  Cultures of skin prior to skin prep are taken to define to native flora at the shoulder and knee area.

CONTACTS AND LOCATIONS:
Overall Officials: Robin M Gehrmann, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ UH, Newark, New Jersey, United States

REFERENCES:
- [Background] Armstrong P, Young C, McKeown D. Ethyl chloride and venepuncture pain: a comparison with intradermal lidocaine. Can J Anaesth. 1990 Sep;37(6):656-8. doi: 10.1007/BF03006485. PMID 2208537
- [Background] Cohen Reis E, Holubkov R. Vapocoolant spray is equally effective as EMLA cream in reducing immunization pain in school-aged children. Pediatrics. 1997 Dec;100(6):E5. doi: 10.1542/peds.100.6.e5. PMID 9374583
- [Background] Soueid A, Richard B. Ethyl chloride as a cryoanalgesic in pediatrics for venipuncture. Pediatr Emerg Care. 2007 Jun;23(6):380-3. doi: 10.1097/01.pec.0000278396.25129.3f. PMID 17572521
- [Background] Weiss JE, Uribe AG, Malleson PN, Kimura Y. Anesthesia for intra-articular corticosteroid injections in juvenile idiopathic arthritis: A survey of pediatric rheumatologists. Pediatr Rheumatol Online J. 2010 Jan 13;8:3. doi: 10.1186/1546-0096-8-3. PMID 20142994
- [Background] Burney K, Bowker K, Reynolds R, Bradley M. Topical ethyl chloride fine spray. Does it have any antimicrobial activity? Clin Radiol. 2006 Dec;61(12):1055-7. doi: 10.1016/j.crad.2006.07.009. PMID 17097428
- [Background] Saltzman MD, Nuber GW, Gryzlo SM, Marecek GS, Koh JL. Efficacy of surgical preparation solutions in shoulder surgery. J Bone Joint Surg Am. 2009 Aug;91(8):1949-53. doi: 10.2106/JBJS.H.00768. PMID 19651954
- [Derived] Polishchuk D, Gehrmann R, Tan V. Skin sterility after application of ethyl chloride spray. J Bone Joint Surg Am. 2012 Jan 18;94(2):118-20. doi: 10.2106/JBJS.K.00229. PMID 22257997